CLINICAL TRIAL: NCT03050606
Title: Effectiveness and Cost-effectiveness of Modified Pilates Method Versus Aerobic Exercise in the Treatment of Patients With Fibromyalgia: a Randomized Controlled Trial
Brief Title: Effectiveness and Cost-effectiveness of Modified Pilates Method Versus Aerobic Exercise in Patients With Fibromyalgia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidade Cidade de Sao Paulo (Other)
Responsible Party: Principal Investigator, Cristina Maria Nunes Cabral, Professor, Universidade Cidade de Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UNICID15
Record Dates: First submitted 2017-02-03; First posted 2017-02-13 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Fibromyalgia
Keywords: Exercise Therapy; Exercise Movement Techniques; Pilates-Based Exercises; Cost-effectiveness
MeSH Terms: conditions — Fibromyalgia | interventions — Exercise Movement Techniques

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pilates (Experimental): This group will perform a modified Pilates exercise program, which will be performed using mat, accessories and studio apparatus, in individual sessions, twice a week, lasting 60 minutes.
  Both groups will also receive an educational booklet with information on fibromyalgia and self-care strategies for pain management, sleep improvement, depression improvement, stress and fatigue control.
  Interventions: Other: Pilates
- Aerobic (Active Comparator): This group will perform aerobic exercise, performed on the treadmill or stationary bike according to the choice of the patient. The training will be performed controlling the heart rate of training. The exercises will be performed individually, twice a week and each session will last 60 minutes.
  Both groups will also receive an educational booklet with information on fibromyalgia and self-care strategies for pain management, sleep improvement, depression improvement, stress and fatigue control.
  Interventions: Other: Aerobic

INTERVENTIONS:
Other: Pilates — Exercises performed on the mat and apparatus, following the six principles of the Pilates method. The exercises will be performed in three levels of difficulty: basic, intermediate and advanced, according to the capacity of the patient.
  Other Names: Modified Pilates method exercises
  Arms: Pilates
Other: Aerobic — Aerobic exercise will be carried out individually on treadmills or stationary bikes. The intensity of the training will be mild to moderate (57% to 76% of the maximal heart rate monitored by the frequencymeter).
  Arms: Aerobic

SUMMARY:
Fibromyalgia is a rheumatologic disease characterized by generalized chronic pain, hyperalgesia and allodynia. Physical exercises are recommended as the first choice of non-pharmacological therapy. Thus, the purpose of this study is to evaluate the effectiveness and cost-effectiveness of modified Pilates method exercises compared to aerobic exercises in the treatment of patients with fibromyalgia. The hypothesis is that Pilates exercises will be as effective as aerobic exercise in the improvement of clinical outcomes, and that this improvement will be maintained over the medium to long term. It is also expected that aerobic exercises will be more cost-effective.

DETAILED DESCRIPTION:
Fibromyalgia is a rheumatologic disease characterized by generalized chronic pain, hyperalgesia and allodynia. Physical exercises are recommended as the first choice of non-pharmacological therapy. Thus, the purpose of this study is to evaluate the effectiveness and cost-effectiveness of modified Pilates method exercises compared to aerobic exercise in the treatment of patients with fibromyalgia. For this, the following outcomes of 98 patients will be evaluated by a blinded evaluator at baseline, 8 weeks, 6 and 12 months after randomization: fibromyalgia impact assessed by the Fibromyalgia Impact Questionnaire, pain intensity assessed by the Pain Numerical Rating Scale, kinesiophobia assessed by the Tampa Scale for Kinesiophobia, specific disability assessed by the Patient-Specific Functional Scale, functional capacity assessed by the 6-minute Walk Test, quality of sleep assessed by the Pittsburgh Sleep Quality Index, and health-related quality of life assessed by the EQ-5D-3L and SF-6D questionnaires. Participants will be randomly divided into Aerobic Group, who will perform aerobic exercises on treadmills and/or stationary bikes, and Pilates Group, which will perform exercises of the modified Pilates method. Both groups will be treated for eight weeks, twice a week. The hypothesis is that Pilates exercises will be as effective as aerobic exercise in the improvement of clinical outcomes, and that this improvement will be maintained over the medium to long term. It is also expected that aerobic exercises will be more cost-effective.

ELIGIBILITY:
Inclusion Criteria:

* Patients that meet the criteria for classification of fibromyalgia according to the criteria of the American College of Rheumatology 2010; and
* Pain intensity greater than or equal to 3 points in the Pain Numerical Rating Scale

Exclusion Criteria:

* Contraindications to physical exercise
* Pregnancy
* Uncontrolled systemic diseases (diabetes mellitus, systemic arterial hypertension and thyroid dysfunctions);
* Neurological, cardiorespiratory and musculoskeletal conditions that interfere with treatment such as: paralysis, significant changes in sensitivity, changes in level of consciousness and understanding, advanced joint diseases (severe arthrosis, hip or knee arthroplasty, severe rheumatoid arthritis), cervicalgia with irradiation to the upper limbs, among others;
* Injury or severe pain in the lower limbs that limit the performance of aerobic exercises: meniscus injury, plantar fasciitis, among others;
* Partial or total muscular ruptures;
* Amputations;
* Recent postoperative; and
* Inability to understand the writing and speaking of the Portuguese language.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2017-02-15 (Actual); Primary Completion 2018-12-22 (Actual); Study Completion 2020-12-22 (Estimated)

PRIMARY OUTCOMES:
Fibromyalgia impact | Eight weeks after randomization
  This outcome will be evaluated by the Fibromyalgia Impact Questionnaire (FIQ) which is composed of 10 items. Item 1 contains 10 questions related to functionality, each of these issues being evaluated by a 4-point Likert scale, which ranges from 0 (always) to 3 (never). In items 2 and 3, the patient scores the number of days that felt well and that was unable to work due to fibromyalgia in the last seven days. Items 4 to 10 are composed of numerical scales that assess difficulty for work, pain, fatigue, morning tiredness, stiffness, anxiety and depression. The FIQ score ranges from 0 to 100 points and the higher values indicate greater fibromyalgia impact on quality of life.

SECONDARY OUTCOMES:
Fibromyalgia impact | Six and twelve months after randomization
  This outcome will be evaluated by the Fibromyalgia Impact Questionnaire (FIQ) which is composed of 10 items. Item 1 contains 10 questions related to functionality, each of these issues being evaluated by a 4-point Likert scale, which ranges from 0 (always) to 3 (never). In items 2 and 3, the patient scores the number of days that felt well and that was unable to work due to fibromyalgia in the last seven days. Items 4 to 10 are composed of numerical scales that assess difficulty for work, pain, fatigue, morning tiredness, stiffness, anxiety and depression. The FIQ score ranges from 0 to 100 points and the higher values indicate greater fibromyalgia impact on quality of life.
Pain intensity | Eight weeks, six and twelve months after randomization
  This outcome will be evaluated by an 11-point scale ranging from 0 to 10, in which 0 represents "no pain" and 10 represents "pain as bad as it could be." The participant will classify his average pain in the last 7days.
Pain intensity | Eigth weeks, before and after each intervention session
  This outcome will be evaluated by an 11-point scale ranging from 0 to 10, in which 0 represents "no pain" and 10 represents "pain as bad as it could be." The participant will classify his average pain before and after each treatment session .
Functional capacity | Eight weeks after randomization
  This outcome will be assessed using the 6-Minute Walk Test. Two cones will be used, which will mark the starting point and 30 meters, where the patient will turn around and continue walking without hesitation. The area of the test will also have markings every 3 meters. The patient should walk for 6 minutes, as fast as he can, without running, while the evaluator will control the time (for 6 minutes) and count how many laps the patient performs (each turn corresponds to 60 meters). When the stopwatch is stopped, the evaluator will say "stop" and mark the point where the patient stopped with a tape. After the test, the evaluator will request that the patient answer to the Borg's range of effort perception. The measurement of the walked distance will be made by the number of laps added to the meters walked until the patient stops.
Kinesiophobia | Eight weeks, six and twelve months after randomization
  This outcome will be evaluated by a 17-item questionnaire. The score of each question varies from 1 ("strongly disagree") to 4 ("strongly agree") points. For the total score, the scores of the questions 4, 8, 12, and 16 should be inverted. The final score can vary from 17 to 68 points, and the higher the score, the greater the degree of kinesiophobia.
Quality of sleep | Eight weeks, six and twelve months after randomization
  This outcome will be evaluated by the Pittsburgh Sleep Quality Index, where the patient will report sleep quality in the last month. The questionnaire consists of 19 self-evaluation questions. The 19 questions are classified into seven components (subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, sleeping medication use and daytime dysfunction), which are rated at a score ranging from 0 to 3 (0 = none in the last month, 1 = less than 1 time/week, 2 = 1 or 2 times/week, 3 = 3 or more times/week). The sum of the scores for these 7 components ranges from 0 to 21, where the highest score indicates poorer sleep quality.
Specific disability | Eight weeks, six and twelve months after randomization
  This outcome will be evaluated using the Patient-Specific Functional Scale. The participants will identify 3 significant activities that are difficult or that are unable to perform because of fibromyalgia. Next, the participants will rate how able they feel to perform these activities on an 11-point scale (0 to 10), with 0 representing "unable to perform activity" and 10 "able to perform the activity at preinjury level." The final score is the mean of the 3 ratings, and the higher the score, the greater the specific ability.
Health-related quality of life using the EQ-5D-3L | Eight weeks, six and twelve months after randomization
  This outcome will be evaluated by the Euroqol 5 dimensions (EQ-5D-3L). The EQ-5D-3L questionnaire is a generic measure that assesses health-related quality of life through five dimensions, and each dimension with three levels. Health states are labeled with a five-digit numeric code that represents the severity level in each dimension.
Health-related quality of life using the SF-6D | Eight weeks, six and twelve months after randomization
  This outcome will be evaluated by the Short-Form 6 dimensions (SF-6D). The SF-6D questionnaire also measures health-related quality of life, through six domains: functional capacity, global limitation, social aspects, pain, mental health and vitality. The SF-6D score represents the strength of an individual's preference for a particular health condition, ranging from zero to one, where zero corresponds to the worst health condition and one corresponds to the best health status.

CONTACTS AND LOCATIONS:
Overall Officials: Cristina MN Cabral, PhD, Principal Investigator — Universidade Cidade de São Paulo
Locations (1):
- Physical Therapy Outpatient Department, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Franco KFM, Miyamoto GC, Franco YRDS, Salvador EMES, do Nascimento BCB, Menten LA, Cabral CMN. Is Pilates more effective and cost-effective than aerobic exercise in the treatment of patients with fibromyalgia syndrome? A randomized controlled trial with economic evaluation. Eur J Pain. 2023 Jan;27(1):54-71. doi: 10.1002/ejp.2039. Epub 2022 Sep 23. PMID 36097826
- [Derived] Franco KFM, Franco YRDS, Salvador EMES, do Nascimento BCB, Miyamoto GC, Cabral CMN. Effectiveness and cost-effectiveness of the modified Pilates method versus aerobic exercise in the treatment of patients with fibromyalgia: protocol for a randomized controlled trial. BMC Rheumatol. 2019 Jan 18;3:2. doi: 10.1186/s41927-018-0051-6. eCollection 2019. PMID 30886990